CLINICAL TRIAL: NCT06794515
Title: Metabolic Effects of cGMP: From Amino Acid Absorption Kinetics to Appetite Modulation
Brief Title: cGMP: Metabolism and Appetite Modulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Nova de Lisboa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: cGMP: Metabolism and Appetite
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — Olive Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Meal A (Experimental): Meal A - CGMP-AAs alone
  Interventions: Dietary Supplement: cGMP-AAs alone (20 g of protein equivalent)
- Meal B (Experimental): Meal B - CGMP-AAs in combination with carbohydrates (including fibre)
  Interventions: Dietary Supplement: cGMP-AAs (20 g of protein equivalent) + 50 g of low-protein bread + 160 g of unpeeled apple
- Meal C (Experimental): Meal C - CGMP-AAs in combination with carbohydrates and fat
  Interventions: Dietary Supplement: cGMP-AAs (20 g of protein equivalent) + 50 g of low-protein bread + 10 g of olive oil

INTERVENTIONS:
Dietary Supplement: cGMP-AAs alone (20 g of protein equivalent) — cGMP-AAs alone (20 g of protein equivalent)
  Arms: Meal A
Dietary Supplement: cGMP-AAs (20 g of protein equivalent) + 50 g of low-protein bread + 160 g of unpeeled apple — cGMP-AAs (20 g of protein equivalent) + 50 g of low-protein bread + 160 g of unpeeled apple
  Arms: Meal B
Dietary Supplement: cGMP-AAs (20 g of protein equivalent) + 50 g of low-protein bread + 10 g of olive oil — cGMP-AAs (20 g of protein equivalent) + 50 g of low-protein bread + 10 g of olive oil
  Arms: Meal C

SUMMARY:
Phenylketonuria is an inborn error of phenylalanine metabolism. Although the phenylalanine-restricted diet is recognized as the mainstay of therapy, little is known about the impact of protein substitutes on the metabolism of patients with phenylketonuria.

Therefore, the aim of this project is to study the impact of acute ingestion of casein glycomacropeptide supplemented with amino acids (cCGMP-AAs) alone or in combination with two different meals on amino acid absorption kinetics, glycaemic and insulinemic response, and on acute markers of appetite control.

The main findings of this project will bring new insights into the dietary management of these patients, which may lead to improvements in protein substitutes formulations.

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* Adults (age ≥ 18 years)
* Body Mass Index (BMI) between 18.5-25.0 kg/m2
* Filling informed consent

Exclusion Criteria:

* Clinically significant illness
* Have changed frequency, duration, or intensity of physical activity in the last month
* Taking protein supplements
* Pregnant or breastfeeding
* Smoking and drug use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-02-03 (Estimated); Primary Completion 2025-03-28 (Estimated); Study Completion 2025-04-24 (Estimated)

PRIMARY OUTCOMES:
Changes in the iAUC (mmol/L*min) for total amino acids | 180 minutes
  Total amino acids will be measured in fasting and every 30 minutes up to 180 minutes. The iAUC (mmol/L*min) for amino acids will be calculated based on the concentration curve following consumption of the test meal.
Changes in the iAUC (pmol/L*min) for glucagon-like peptide-1 (GLP-1) | 180 minutes
  GLP-1 will be measured in fasting and every 30 minutes up to 180 minutes. The iAUC (pmol/L*min) for GLP-1 will be calculated based on the concentration curve following consumption of the test meal.
Changes in the iAUC (pmol/L*min) for Cholecystokinin (CCK) | 180 minutes
  CCK will be measured in fasting and every 30 minutes up to 180 minutes. The iAUC (pmol/L*min) for CCK will be calculated based on the concentration curve following consumption of the test meal.
Changes in the iAUC (pmol/L*min) for peptide YY (PYY) | 180 minutes
  PYY will be measured in fasting and every 30 minutes up to 180 minutes. The iAUC (pmol/L*min) for PYY will be calculated based on the concentration curve following consumption of the test meal.
Changes in the iAUC (pmol/L*min) for Gastric inhibitory polypeptide (GIP) | 180 minutes
  GIP will be measured in fasting and every 30 minutes up to 180 minutes. The iAUC (pmol/L*min) for GIP will be calculated based on the concentration curve following consumption of the test meal.

SECONDARY OUTCOMES:
Changes in glucose | 180 minutes
  Glucose will be measured in fasting and every 30 minutes up to 3 hours. The iAUC (mmol/L*min) for glucose will be calculated based on the concentration curve following consumption of the test meal.
Changes in insulin | 180 minutes
  Insulin will be measured in fasting and every 30 minutes up to 3 hours. The iAUC (mmol/L*min) for insulin will be calculated based on the concentration curve following consumption of the test meal.
Changes in C-peptide | 180 minutes
  C-peptide will be measured in fasting and every 30 minutes up to 3 hours. The iAUC (mmol/L*min) for C-peptide will be calculated based on the concentration curve following consumption of the test meal.

CONTACTS AND LOCATIONS:
Locations (1):
- NOVA Medical School|Faculdade de Ciências Médicas, Universidade NOVA de Lisboa, Lisboa,, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No